CLINICAL TRIAL: NCT06805877
Title: Predictive Analytics and Clinical Decision Support to Improve PrEP Prescribing in Community Health Centers
Brief Title: Predictive Analytics and Clinical Decision Support to Improve PrEP Prescribing
Acronym: PrEDICT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); OCHIN, Inc. (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Julia Marcus, Associate Professor, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PH001008; R01MH133515 (NIH)
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: HIV
Keywords: HIV; PrEP; pre-exposure prophylaxis; prevention; prediction model; clinical decision support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Data will be extracted from EHRs of control clinics as a comparison, and those clinics will not actively participate in study activities
- Predictive analytics and clinical decision support (Active Comparator): Providers in enrolled intervention clinics will receive point-of-care notifications via the EHR-embedded decision support tool about patients who are at increased predicted HIV risk and therefore likely to benefit from PrEP
  Interventions: Other: Predictive Analytics and Clinical Decision Support

INTERVENTIONS:
Other: Predictive Analytics and Clinical Decision Support — The intervention will include automated EHR notifications to clinicians at 16 OCHIN community health centers about patients who are likely to benefit from PrEP. These patients will be identified by an HIV prediction model that was developed and validated during the pilot phase of this study using historical OCHIN EHR data. For patients above a preselected threshold of predicted HIV risk, clinicians will be notified at the point of care that the patient may benefit from PrEP and will be provided with EHR-based tools to support discussions and prescribing. The intervention will also include coaching on PrEP and the decision support tool, as well as project team support during the trial period.
  Arms: Predictive analytics and clinical decision support

SUMMARY:
Scale-up of HIV preexposure prophylaxis (PrEP) is a key strategy of the U.S. initiative to end the HIV epidemic, but healthcare providers lack tools to support PrEP discussions and prescribing for patients likely to benefit. This research will evaluate whether integrating automated tools into electronic health records to help providers efficiently and equitably identify potential candidates for PrEP, discuss PrEP, and prescribe PrEP can improve PrEP initiation and persistence in safety-net community health centers. It will achieve this by conducting a stepped-wedge trial of a decision support tool with an embedded HIV prediction model to identify patients likely to benefit from PrEP. The intervention will be delivered to healthcare providers in 16 community health centers within the national OCHIN network.

ELIGIBILITY:
Inclusion Criteria:

* Delivery site saw at least 500 distinct patients in 2024 during in-person or telehealth visits
* Delivery site had at least 10 new HIV diagnoses or positive HIV screening tests in 2023
* Delivery site provides primary care other than pediatrics, and the primary care department(s) were active on OCHIN Epic as of 1/1/2023

Exclusion Criteria:

* Delivery site specializing in HIV or STI care
* Correctional facilities
* Mobile sites
* School-based health center sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
PrEP initation | 30 months
  Proportion of patients above the prediction model risk threshold without a recently active PrEP prescription (within the prior 6 months) or prior HIV diagnosis who are prescribed PrEP during the study period.

SECONDARY OUTCOMES:
PrEP persistence | 30 months
  Proportion of patients prescribed PrEP who persist on PrEP for 6 and 12 months, as measured by prescription refills ordered.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Bay Area Community Health Liberty Clinic, Fremont, California
  - Lifelong East Oakland Health Center, Oakland, California
  - TrueCare Oceanside Family Medicine, Oceanside, California
  - DAP Legacy, Palm Springs, California
  - One Community Health Midtown Campus, Sacramento, California
  - Southwest Community Health Center 968 Fairfield Avenue, Bridgeport, Connecticut
  - Mercy Care Decatur Street, Atlanta, Georgia
  - Siouxland Community Health Center Sioux City, Sioux City, Iowa
  - Lynn Community Health Center 269 Union, Lynn, Massachusetts
  - Mattapan Community Health Center Blue Hill, Mattapan, Massachusetts
  - Neighborhood Family Practice Ridge Community Health Center, Cleveland, Ohio
  - Signature Health Painesville, Painesville, Ohio
  - Variety Care Sequoyah, Oklahoma City, Oklahoma
  - Prism Belmont, Portland, Oregon
  - Bee Busy Wellness Center Bray Oaks, Houston, Texas
  - Seattle Roots Community Health Carolyn Downs Community Clinic, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No